CLINICAL TRIAL: NCT05462587
Title: A Phase 3, Randomized, Double-blind, Two-period, Crossover, Withdrawal Study to Assess the Efficacy and Safety of AVTX-803 in Subjects with Leukocyte Adhesion Deficiency Type II (LAD II)
Brief Title: A Study to Evaluate Efficacy and Safety of AVTX-803 in Patients with Leukocyte Adhesion Deficiency Type II
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AUG Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: AVTX-803-LAD-301
Record Dates: First submitted 2022-06-28; First posted 2022-07-18 (Actual); Last update posted 2024-11-01 (Actual); Status verified 2024-03

CONDITIONS: Leukocyte Adhesion Deficiency
MeSH Terms: conditions — Leukocyte adhesion deficiency type 1 | interventions — Fucose

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- AVTX-803 (Experimental): Approximately 4 subjects will receive AVTX-803 at a dose specified by the investigator up to 5 times a day not to exceed 1700 mg/kg/day for 8 weeks.
  Interventions: Drug: AVTX-803 (L-Fucose)
- Withdrawal (No Intervention): Subject will be in withdrawal for 8 weeks.

INTERVENTIONS:
Drug: AVTX-803 (L-Fucose) — L-fucose crystalline powder
  Arms: AVTX-803

SUMMARY:
The primary objective of this study is to evaluate the efficacy and safety of AVTX-803 compared to withdrawal in patients with Leukocyte Adhesion Deficiency, Type II (LAD II).

ELIGIBILITY:
Inclusion Criteria:

* Subject must be between 6 months and 75 years old
* Subject has biochemically and genetically proven LAD II (SLC35C1-CDG)
* Subject has a documented history of Lewis antigen deficiency
* Subject has a history of recurrent infections, opportunistic infections or infections that did not respond well to standard of care treatment
* Subject or parent (for subjects under legal age for consent) has provided written informed consent for this study. Additionally, written informed assent has been provided, as appropriate, for minors of older age, per local institutional review board (IRB)/ethics committee (EC) policy and requirements
* Subject is willing and able to comply with the protocol
* Women of childbearing potential (WOCBP) meeting the criteria below:

  1. Non-lactating and has a negative pregnancy test at screening -AND-
  2. Uses an acceptable double-barrier method of contraception as determined by the investigator or sub-investigator for the duration of the study and 30 days following the last dose of study drug.
* Male subjects must agree to use an acceptable double-barrier method of contraception with their partner as determined by the investigator or sub-investigator for the duration of the study and 30 days following the last dose of study drug.

Exclusion Criteria:

* Subject has severe anemia defined as hemoglobin <8.0 g/dL (<4.9 mmol/L)
* Subject has impaired renal function as defined by an eGFR <90 mL/min
* Subject has a total absence of fucosylation on red blood cells and the presence of anti-H antigen
* Subject has known or suspected intolerance or hypersensitivity to fucose or any ingredients of the investigational product
* In the investigator's opinion, subject has a history of failure to respond to fucose at adequate dosing
* In the investigator's opinion, subject is not able or not willing to comply with the study requirements.
* Subject is pregnant

Ages: 6 Months to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 4 (Estimated)
Dates: Start 2022-07-28 (Actual); Primary Completion 2024-11-30 (Estimated); Study Completion 2024-11-30 (Estimated)

PRIMARY OUTCOMES:
Effect of AVTX-803 on the percent of leukocytes expressing Sialyl-Lewis X antigen | Change from Baseline at Day 56, Change from Baseline at Day 112
  To assess the effect of AVTX-803 in subjects with leukocyte adhesion deficiency Type II (LAD II) by evaluating Sialyl-Lewis X on leukocytes as a percentage present at the end of each 8 week treatment period.

CONTACTS AND LOCATIONS:
Overall Officials: David Deyle, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No